CLINICAL TRIAL: NCT00404911
Title: Family Groups to Reduce Youth Behavioral Difficulties
Brief Title: Multi-Family Group Therapy for Reducing Behavioral Difficulties in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 04-0063; R01MH072649 (NIH); DSIR CT-C
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Oppositional Defiant Disorder; Conduct Disorder
Keywords: Oppositional Defiant Disorder
MeSH Terms: conditions — Oppositional Defiant Disorder; Conduct Disorder | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MFG therapy (Experimental): Participants will receive multi-family group therapy
  Interventions: Behavioral: MFG therapy; Behavioral: Standard of Care
- Standard of Care (Active Comparator): Participants will receive standard care
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: MFG therapy — MFG includes 16 weekly group therapy sessions for families with children who have ODD or CD. Sessions will include adult caregivers and all children over age 6. Each session will follow the same procedures, and will proceed through the following stages: creating social networks; information exchange; group discussions; individual family practice; and homework assignment.
  Other Names: Multiple Family Group Project
  Arms: MFG therapy
Behavioral: Standard of Care — Participants assigned to standard care will receive treatment that is traditionally offered to outpatients. Participants in the MFG program will also receive standard care.
  Other Names: Multiple Family Group Project; Standard care control

SUMMARY:
This study will examine the effectiveness of a multiple family group mental health service delivery strategy in improving mental health service use and outcome for urban, low income children of color, ages 7-11 years old with disruptive behaviors and their families.

DETAILED DESCRIPTION:
Oppositional defiant disorder (ODD) and conduct disorder (CD) are two common childhood psychiatric disorders. Children with ODD frequently have temper tantrums, argue excessively with adults, deliberately attempt to annoy or upset people, and blame others for their mistakes or behavior. Children with CD may exhibit aggression toward people and animals, destruction of property, deceitfulness, and rule breaking. The symptoms of these disorders can negatively affect children's social, family, and academic lives. Research has shown that early, comprehensive treatment leads to better treatment outcomes. Both disorders are commonly treated using parent training techniques. A multiple family group therapy setting may prove to be more engaging and beneficial than standard care for both parents and children. This study will examine the effectiveness of a multiple family group (MFG) mental health service delivery strategy in improving mental health service use and treatment outcome for urban, low income children of color with ODD or CD.

Participants in this 18-month, open-label study will be randomly assigned to either receive standard of care or participate in an MFG in addition to receiving standard of care. Participants assigned to standard of care will receive treatment that is traditionally offered to outpatients. Participants in an MFG will meet in their groups once a week for 16 weeks. Sessions will include adult caregivers and all children over age 6. Each session will follow the same procedures, and will proceed through the following stages: creating social networks; information exchange; group discussions; individual family practice; and homework assignment. Assessments of youth functioning will be held at Weeks 8 and 16 and Months 6 and 18 post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Youth participants are between the ages of 7 and 11
* Adult caregivers are available to participate in the research and intervention activities
* Both youth and adult caregiver are English- or Spanish-speaking
* Youth meets criteria for a primary diagnosis of oppositional defiant disorder or conduct disorder, as measured by the Disruptive Behavior Disorder Rating Scale (DBD)

Exclusion Criteria:

* Youth has significant cognitive impairment that might interfere with understanding of program content or informed consent process
* Youth or adult has emergency psychiatric needs that require services beyond those provided within an outpatient setting (e.g., hospitalization or specialized placement outside the home)
* Youth who are wards of the state

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2006-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Youth externalizing behaviors and functioning | Measured at week 16 of treatment
Youth externalizing behaviors and functioning | Measured 6 Months follow-up visit

SECONDARY OUTCOMES:
Parenting skills | 16 weeks and 6 months
  change in parenting skills after intervention
Involvement in child mental health care | 16 weeks and 6 months
  comparison of involvement in child mental health care after intervention
Parent/child interaction | 16 weeks and 6 months
  change in parent and child interaction after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mary M. McKay, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai, Department of Psychiatry
Locations (1):
- Mount Sinai's Child and Adolescent Outpatient Psychiatry Clinic, New York, New York, United States